CLINICAL TRIAL: NCT02500888
Title: Initial Evaluation of Efficacy and Adverse Events of Single Lesions in Bilateral Ventral-capsular and Ventral Capsulotomy-striatal by Linear Accelerator Radiosurgery in Severe and Refractory Obsessive-compulsive Disorder
Brief Title: Evaluation of Capsulotomy by Linear Accelerator Radiosurgery in Severe and Refractory Obsessive-compulsive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-0341
Record Dates: First submitted 2015-07-09; First posted 2015-07-17 (Estimated); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: OCD; Quality of Life
Keywords: OCD; Neurosurgery; Radiosurgery
MeSH Terms: interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Radiosurgery by linear accelerator.
  Interventions: Radiation: Radiosurgery

INTERVENTIONS:
Radiation: Radiosurgery — Only one radiation session of about 180 Gy in bilateral internal capsule.

SUMMARY:
The aim of this study is to evaluate, through a pilot study with about ten cases, if bilateral ventral capsulotomy by linear accelerator enable modification of obsessive-compulsive symptoms and quality of life in patients with severe and refractory obsessive compulsive disorder (OCD) and also investigate possible adverse effects / complications of the procedure.

DETAILED DESCRIPTION:
About ten patients with severe and refractory OCD will receive bilateral single lesions at the bottom of the anterior limb of the internal capsule by linear accelerator. Prior to the procedure, a detailed clinical and psychiatric evaluation, plus an extensive battery of psychiatric diagnostic tests, severity and progression of OCD, depression / anxiety symptoms, presence of tics, psychosocial impairment, quality of life, familial accommodation and neuropsychological and personality testes will be performed. Furthermore, the patients will be also assessed by serological and neuroimaging tests. The Individuals will be periodically evaluated and followed up for one year. The results of the scores of the rating scales will be analyzed and compared, as well as the profile of adverse events, cognitive or personality changes and improves in clinical tests and neuroimaging studies.

ELIGIBILITY:
Inclusion Criteria:

1. OCD diagnosis, according to Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) as a major disease entity. If comorbidity with other psychiatric or personality disorders, OCD symptoms dominate the clinical picture and precede other disorders.
2. Duration of OCD symptoms of at least five years.
3. Scores range of the obsessive-compulsive symptoms "Yale-Brown Obsessive-Compulsive Scale" (YBOCS) greater than 26 (or greater than 13, if obsessions or compulsions alone).
4. Fill up the criteria for refractory to prior treatments.
5. Be accepted by the method of "best estimate" for defining the patient is refractory, which consisted of confirmation by at least two specialists obsessive-compulsive disorder that the patient fulfills the criteria for effective refractory to previous treatments.

Exclusion Criteria:

1. History of head trauma or post-traumatic amnesia.
2. Background of systemic or neurological diseases with brain impairment, severe and active.
3. History of current use of substances capable of inducing psychopathological manifestations, or signs of cumulative effects of alcohol or drugs in the central nervous system (such as cortical atrophy), confirmed by neuroimaging.
4. pregnancy or lactation.
5. Refusal to submit to the radiosurgical procedure.
6. Refusal to accept the informed consent form, or participate.
7. History of mental retardation and / or inability to understand the informed consent, confirmed by neuropsychological tests of the initial evaluation.
8. Lack of family or companion with proper capacity of understanding of the informed consent in patients with comorbid major depression or psychosis that could potentially have difficulty performing the appropriate judgment as to participate in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2015-06-30 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in OCD symptoms | Every 3 months until 12 months
  Application of Yale-Brown Obsessive-Compulsive Scale (Y-Bocs) scale

SECONDARY OUTCOMES:
Change in quality of life. | Every 3 months until 12 months
  Application of "Medical Outcomes Study 36-Item Short-Form Health Survey" (SF-36) scale
Change in brain-derived neurotrophic factor (BDNF) blood dosing | 12 months
  Serological blood tests
Change in psychological tests | 12 months
  Application of:
  * Mini Mental Modified (3MS) test
  * Wechsler of intelligence test
  * Stroop of colors test
  * Tracks tests A and B
  * Boston Naming Test (BNT)
  * Wechsler Memory Scale Revised (WMS-R)
  * Wisconsin (WCST) test
  * Brief Visual Memory Test (BVLT)
  * Hopkins Verbal Learning Test (HBLT) test
  * Benton Line Orientation (BLO) test
  * Grooved Pegboard Test
  * Finger Tapping test
  * Complex figure of Rey test
Side effects and complications | Every 3 months until 12 months
  Application of "Systematic Assessment for Treatment Emergent Effects" (SAFTEE) Event List and Interview.
Change in familial accommodation | Every 3 months until 12 months
  Application of "Family Accommodation Scale for Obsessive-Compulsive Disorder" (FAS)
Change in anxiety symptoms. | Every 3 months until 12 months
  Application of "Beck Anxiety Inventory" (BAI) scale
Change in depressive symptoms. | Every 3 months until 12 months
  Application of "Beck Depression Inventory" (BDI) scale
Change in near-infrared spectroscopy (NIRS) brain blood flow | 12 months
  During application of Stroop psychological test.
Change in OCD symptoms by CPRS | Every 3 months
  Application of "Comprehensive Psychopathological Rating Scale" (CPRS)
Change in OCD symptoms by NIMH. | Every 3 months
  Application of "National Institute of Mental Health Global Obsessive-Compulsive Scale" (NIMH OCD Scale)
Change in Global Functioning | Every 3 months until 12 months
  Application of "Global Assessment of Functioning Scale" (GAF)

CONTACTS AND LOCATIONS:
Overall Officials: Paulo Abreu, M.D.; Ph.D., Principal Investigator — Professor of Medicine
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Asberg M, Montgomery SA, Perris C, Schalling D, Sedvall G. A comprehensive psychopathological rating scale. Acta Psychiatr Scand Suppl. 1978;(271):5-27. doi: 10.1111/j.1600-0447.1978.tb02357.x. No abstract available. PMID 277059
- [Background] Ballantine HT Jr, Cassidy WL, Flanagan NB, Marino R Jr. Stereotaxic anterior cingulotomy for neuropsychiatric illness and intractable pain. J Neurosurg. 1967 May;26(5):488-95. doi: 10.3171/jns.1967.26.5.0488. No abstract available. PMID 5337782
- [Background] Batistuzzo MC, Taub A, Nakano E, D'Alcante CC, de Mathis ME, Hoexter MQ, Miguel EC, Lopes AC. Performance of patients with refractory obsessive-compulsive disorder in the Frontal Systems Behavior Scale. Neurocase. 2009;15(2):157-62. doi: 10.1080/13554790802709047. Epub 2009 Mar 9. PMID 19274575
- [Background] Beck AT, Epstein N, Brown G, Steer RA. An inventory for measuring clinical anxiety: psychometric properties. J Consult Clin Psychol. 1988 Dec;56(6):893-7. doi: 10.1037//0022-006x.56.6.893. No abstract available. PMID 3204199
- [Background] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369
- [Background] Brandt RA, Salvajoli JV, Oliveira VC, Carmignani M, da Cruz JC, Leal HD, Ferraz L. [Linear accelerator radiosurgery]. Arq Neuropsiquiatr. 1995 Mar;53(1):38-45. doi: 10.1590/s0004-282x1995000100007. Portuguese. PMID 7575207
- [Background] Calvocoressi L, Libman D, Vegso SJ, McDougle CJ, Price LH. Global functioning of inpatients with obsessive-compulsive disorder, schizophrenia, and major depression. Psychiatr Serv. 1998 Mar;49(3):379-81. doi: 10.1176/ps.49.3.379. PMID 9525801
- [Background] Calvocoressi L, Mazure CM, Kasl SV, Skolnick J, Fisk D, Vegso SJ, Van Noppen BL, Price LH. Family accommodation of obsessive-compulsive symptoms: instrument development and assessment of family behavior. J Nerv Ment Dis. 1999 Oct;187(10):636-42. doi: 10.1097/00005053-199910000-00008. PMID 10535658
- [Background] Cecconi JP, Lopes AC, Duran FL, Santos LC, Hoexter MQ, Gentil AF, Canteras MM, Castro CC, Noren G, Greenberg BD, Rauch SL, Busatto GF, Miguel EC. Gamma ventral capsulotomy for treatment of resistant obsessive-compulsive disorder: a structural MRI pilot prospective study. Neurosci Lett. 2008 Dec 12;447(2-3):138-42. doi: 10.1016/j.neulet.2008.09.061. Epub 2008 Sep 27. PMID 18835422
- [Background] Fodstad H, Strandman E, Karlsson B, West KA. Treatment of chronic obsessive compulsive states with stereotactic anterior capsulotomy or cingulotomy. Acta Neurochir (Wien). 1982;62(1-2):1-23. doi: 10.1007/BF01402207. PMID 7048859
- [Background] Frighetto L, De Salles A, Wallace R, Ford J, Selch M, Cabatan-Awang C, Solberg T. Linear accelerator thalamotomy. Surg Neurol. 2004 Aug;62(2):106-13; discussion 113-4. doi: 10.1016/j.surneu.2003.08.033. PMID 15261496
- [Background] Frighetto L, Bizzi J, Annes RD, Silva Rdos S, Oppitz P. Stereotactic radiosurgery for movement disorders. Surg Neurol Int. 2012;3(Suppl 1):S10-6. doi: 10.4103/2152-7806.91605. Epub 2012 Jan 14. PMID 22826805
- [Background] Goodman WK, Price LH, Rasmussen SA, Mazure C, Delgado P, Heninger GR, Charney DS. The Yale-Brown Obsessive Compulsive Scale. II. Validity. Arch Gen Psychiatry. 1989 Nov;46(11):1012-6. doi: 10.1001/archpsyc.1989.01810110054008. PMID 2510699
- [Background] Lopes AC, Greenberg BD, Canteras MM, Batistuzzo MC, Hoexter MQ, Gentil AF, Pereira CA, Joaquim MA, de Mathis ME, D'Alcante CC, Taub A, de Castro DG, Tokeshi L, Sampaio LA, Leite CC, Shavitt RG, Diniz JB, Busatto G, Noren G, Rasmussen SA, Miguel EC. Gamma ventral capsulotomy for obsessive-compulsive disorder: a randomized clinical trial. JAMA Psychiatry. 2014 Sep;71(9):1066-76. doi: 10.1001/jamapsychiatry.2014.1193. PMID 25054836
- [Background] Guy W, Wilson WH, Brooking B, Manov G, Fjetland O. Reliability and validity of SAFTEE: preliminar analyses. Psychopharmacol Bull. 1986;22(2):397-401. No abstract available. PMID 3774933
- [Background] Hou J, Wu W, Lin Y, Wang J, Zhou D, Guo J, Gu S, He M, Ahmed S, Hu J, Qu W, Li H. Localization of cerebral functional deficits in patients with obsessive-compulsive disorder: a resting-state fMRI study. J Affect Disord. 2012 May;138(3):313-21. doi: 10.1016/j.jad.2012.01.022. Epub 2012 Feb 12. PMID 22331021
- [Background] Huang EJ, Reichardt LF. Neurotrophins: roles in neuronal development and function. Annu Rev Neurosci. 2001;24:677-736. doi: 10.1146/annurev.neuro.24.1.677. PMID 11520916
- [Background] Jenike MA, Rauch SL. Managing the patient with treatment-resistant obsessive compulsive disorder: current strategies. J Clin Psychiatry. 1994 Mar;55 Suppl:11-7. PMID 7915709
- [Background] Kelly DH, Walter CJ, Sargant W. Modified leucotomy assessed by forearm blood flow and other measurements. Br J Psychiatry. 1966 Sep;112(490):871-81. doi: 10.1192/bjp.112.490.871. No abstract available. PMID 5970906
- [Background] KNIGHT G. THE ORBITAL CORTEX AS AN OBJECTIVE IN THE SURGICAL TREATMENT OF MENTAL ILLNESS. THE RESULTS OF 450 CASES OF OPEN OPERATION AND THE DEVELOPMENT OF THE STEREOTACTIC APPROACH. Br J Surg. 1964 Feb;51:114-24. doi: 10.1002/bjs.1800510207. No abstract available. PMID 14117767
- [Background] Leckman JF, Riddle MA, Hardin MT, Ort SI, Swartz KL, Stevenson J, Cohen DJ. The Yale Global Tic Severity Scale: initial testing of a clinician-rated scale of tic severity. J Am Acad Child Adolesc Psychiatry. 1989 Jul;28(4):566-73. doi: 10.1097/00004583-198907000-00015. PMID 2768151
- [Background] Leveque M, Carron R, Regis J. Radiosurgery for the treatment of psychiatric disorders: a review. World Neurosurg. 2013 Sep-Oct;80(3-4):S32.e1-9. doi: 10.1016/j.wneu.2013.07.004. Epub 2013 Jul 17. PMID 23872618
- [Background] Lippitz B, Mindus P, Meyerson BA, Kihlstrom L, Lindquist C. Obsessive compulsive disorder and the right hemisphere: topographic analysis of lesions after anterior capsulotomy performed with thermocoagulation. Acta Neurochir Suppl. 1997;68:61-3. doi: 10.1007/978-3-7091-6513-3_11. PMID 9233415
- [Background] McDougle CJ, Goodman WK, Leckman JF, Lee NC, Heninger GR, Price LH. Haloperidol addition in fluvoxamine-refractory obsessive-compulsive disorder. A double-blind, placebo-controlled study in patients with and without tics. Arch Gen Psychiatry. 1994 Apr;51(4):302-8. doi: 10.1001/archpsyc.1994.03950040046006. PMID 8161290
- [Background] Miguel EC, Coffey BJ, Baer L, Savage CR, Rauch SL, Jenike MA. Phenomenology of intentional repetitive behaviors in obsessive-compulsive disorder and Tourette's disorder. J Clin Psychiatry. 1995 Jun;56(6):246-55. PMID 7775367
- [Background] Mindus P, Rasmussen SA, Lindquist C. Neurosurgical treatment for refractory obsessive-compulsive disorder: implications for understanding frontal lobe function. J Neuropsychiatry Clin Neurosci. 1994 Fall;6(4):467-77. doi: 10.1176/jnp.6.4.467. PMID 7841817
- [Background] Myers JK, Weissman MM, Tischler GL, Holzer CE 3rd, Leaf PJ, Orvaschel H, Anthony JC, Boyd JH, Burke JD Jr, Kramer M, et al. Six-month prevalence of psychiatric disorders in three communities 1980 to 1982. Arch Gen Psychiatry. 1984 Oct;41(10):959-67. doi: 10.1001/archpsyc.1984.01790210041006. PMID 6332591
- [Background] Okada K, Ota T, Iida J, Kishimoto N, Kishimoto T. Lower prefrontal activity in adults with obsessive-compulsive disorder as measured by near-infrared spectroscopy. Prog Neuropsychopharmacol Biol Psychiatry. 2013 Jun 3;43:7-13. doi: 10.1016/j.pnpbp.2012.11.013. Epub 2012 Dec 5. PMID 23220093
- [Background] Ota T, Iida J, Sawada M, Suehiro Y, Yamamuro K, Matsuura H, Tanaka S, Kishimoto N, Negoro H, Kishimoto T. Reduced prefrontal hemodynamic response in pediatric obsessive-compulsive disorder as measured by near-infrared spectroscopy. Child Psychiatry Hum Dev. 2013 Apr;44(2):265-77. doi: 10.1007/s10578-012-0323-0. PMID 22833309
- [Background] Perse T. Obsessive-compulsive disorder: a treatment review. J Clin Psychiatry. 1988 Feb;49(2):48-55. PMID 2892831
- [Background] Rasmussen SA, Eisen JL. Treatment strategies for chronic and refractory obsessive-compulsive disorder. J Clin Psychiatry. 1997;58 Suppl 13:9-13. PMID 9402914
- [Background] Robins LN, Helzer JE, Weissman MM, Orvaschel H, Gruenberg E, Burke JD Jr, Regier DA. Lifetime prevalence of specific psychiatric disorders in three sites. Arch Gen Psychiatry. 1984 Oct;41(10):949-58. doi: 10.1001/archpsyc.1984.01790210031005. PMID 6332590
- [Background] Rylander G. [Experiments with gammacapsulotomy in anxiety and compulsive neuroses]. Lakartidningen. 1978 Feb 15;75(7):547-9. No abstract available. Swedish. PMID 342844
- [Background] Spiegel EA, Wycis HT, Marks M, Lee AJ. Stereotaxic Apparatus for Operations on the Human Brain. Science. 1947 Oct 10;106(2754):349-50. doi: 10.1126/science.106.2754.349. No abstract available. PMID 17777432
- [Background] Steketee G. Disability and family burden in obsessive-compulsive disorder. Can J Psychiatry. 1997 Nov;42(9):919-28. doi: 10.1177/070674379704200902. PMID 9429061
- [Background] Wang Y, Mathews CA, Li Y, Lin Z, Xiao Z. Brain-derived neurotrophic factor (BDNF) plasma levels in drug-naive OCD patients are lower than those in healthy people, but are not lower than those in drug-treated OCD patients. J Affect Disord. 2011 Sep;133(1-2):305-10. doi: 10.1016/j.jad.2011.04.002. Epub 2011 May 25. PMID 21616543
- [Background] Ware JE Jr, Kosinski M, Bayliss MS, McHorney CA, Rogers WH, Raczek A. Comparison of methods for the scoring and statistical analysis of SF-36 health profile and summary measures: summary of results from the Medical Outcomes Study. Med Care. 1995 Apr;33(4 Suppl):AS264-79. PMID 7723455